CLINICAL TRIAL: NCT00428935
Title: Phase 1 Clinical Trial of rAAV2.5-CMV-mini-Dystrophin Gene Vector in Duchenne Muscular Dystrophy
Brief Title: Safety Study of Mini-dystrophin Gene to Treat Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: AskBio Inc (Industry)
Responsible Party: Principal Investigator, Jerry R. Mendell, Director Center for Gene Therapy, Nationwide Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCRI IRB05-00118
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; Muscle; Muscular Dystrophy; Gene Therapy; Dystrophin; Adeno-Associated Virus; AAV
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Low Dose (Experimental): Low dose cohort - 2.0E10 vg/kg
  Interventions: Biological: rAAV2.5-CMV-minidystrophin (d3990)
- High Dose (Experimental): High Dose - 1.0E11 vg/kg
  Interventions: Biological: rAAV2.5-CMV-minidystrophin (d3990)

INTERVENTIONS:
Biological: rAAV2.5-CMV-minidystrophin (d3990) — Recombinant adeno-associated virus (AAV) carrying a truncated human dystrophin gene (mini-dystrophin) expressed from a cytomegalovirus (CMV) promoter.

SUMMARY:
The purpose of this study is to determine the safety of a miniature dystrophin gene in the treatment of progressive muscle weakness due to Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
This phase I randomized double blind dose escalation study investigates the safety and efficacy of the mini-dystrophin gene transferred to the biceps muscle for Duchenne muscular dystrophy patients, ages 5 to 12 years of age, using a recombinant adeno-associated virus. Eligible participants must have a known dystrophin gene mutation and may be concurrently treated with corticoid steroids. The mini-dystrophin gene or a placebo agent (normal saline or empty viral capsids) are injected directly into both biceps muscles while under conscious sedation. Following the gene transfer, patients are admitted to the hospital for 48 hours of observation followed by weekly outpatient visits at the Columbus Children's Hospital Neuromuscular Clinic. A bilateral muscle biopsy is preformed following 6 weeks with long term follow up will consisting of bi-annual visits for the next 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Known null mutation of the Dystrophin gene
* Male age of 5 years or older
* If taking corticosteroids, must have dose unchanged for the past 3 months
* Serum creatine kinase elevation greater than 10x normal value (established by Children's Hospital)
* Progressive, symmetrical proximal muscle weakness of arms and legs

Exclusion Criteria:

* Unable to cooperate for muscle strength testing
* Joint contractures that prohibit muscle strength testing
* Concomitant illness
* Individuals predisposed to excessive vagal responses (bradyarrhythmia or hypotension)
* Controlled substance abuse

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | followed for 2 years post injection
  Physical Exams assessing major organ systems and safety labs (GGT, Bilirubin, Glucose, Amylase, CBC/Diff, AFP, Platelets, PT/PTT, Creatinine, Electrolytes, Total protein, Alkaline phosphatase, and Urinalysis)

SECONDARY OUTCOMES:
mini-dystrophin gene expression at the site of gene transfer | 90 days post injection
Maximal Volume Isometric Contraction Testing as a measure of muscle strength | out to 2 years post injection

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Columbus Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Watchko J, O'Day T, Wang B, Zhou L, Tang Y, Li J, Xiao X. Adeno-associated virus vector-mediated minidystrophin gene therapy improves dystrophic muscle contractile function in mdx mice. Hum Gene Ther. 2002 Aug 10;13(12):1451-60. doi: 10.1089/10430340260185085. PMID 12215266
- [Background] Wang B, Li J, Xiao X. Adeno-associated virus vector carrying human minidystrophin genes effectively ameliorates muscular dystrophy in mdx mouse model. Proc Natl Acad Sci U S A. 2000 Dec 5;97(25):13714-9. doi: 10.1073/pnas.240335297. PMID 11095710
- [Result] Mendell JR, Campbell K, Rodino-Klapac L, Sahenk Z, Shilling C, Lewis S, Bowles D, Gray S, Li C, Galloway G, Malik V, Coley B, Clark KR, Li J, Xiao X, Samulski J, McPhee SW, Samulski RJ, Walker CM. Dystrophin immunity in Duchenne's muscular dystrophy. N Engl J Med. 2010 Oct 7;363(15):1429-37. doi: 10.1056/NEJMoa1000228. PMID 20925545
- [Result] Bowles DE, McPhee SW, Li C, Gray SJ, Samulski JJ, Camp AS, Li J, Wang B, Monahan PE, Rabinowitz JE, Grieger JC, Govindasamy L, Agbandje-McKenna M, Xiao X, Samulski RJ. Phase 1 gene therapy for Duchenne muscular dystrophy using a translational optimized AAV vector. Mol Ther. 2012 Feb;20(2):443-55. doi: 10.1038/mt.2011.237. Epub 2011 Nov 8. PMID 22068425
- See also: Columbus Children's Research Institute — http://www.ccri.net
- See also: Asklepios BioPharmaceutical Inc. — http://www.askbio.com
- See also: Muscular Dystrophy Association — http://www.mdausa.org